CLINICAL TRIAL: NCT02335944
Title: A Phase Ib/II, Multicenter, Open-label Study of EGF816 in Combination With INC280 in Adult Patients With EGFR Mutated Non-small Cell Lung Cancer.
Brief Title: Study of Safety and Efficacy of EGFR-TKI EGF816 in Combination With cMET Inhibitor INC280 in Adult Patients With EGFR Mutated Non Small Cell Lung Cancer.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2105C; 2014-000726-37 (EudraCT Number)
Record Dates: First submitted 2014-10-09; First posted 2015-01-12 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; NSCLC; EGF816; INC280; tyrosine kinase inhibitor; c-MET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib; nazartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase IB part- NSCLC with EGFR activating mutations (Experimental): NSCLC participants who have previously documented EGFR mutation and progressed on EGFR TKI treatment. Participants were treated at a starting dose of 50 mg once a day for EGF816 and 200 mg twice a day for INC280 in fasted state
  Interventions: Drug: Capmatinib; Drug: Nazartinib
- Phase II- Group 1 (EGFRmut, any T790M, any MET, 2/4L antineoplastic, EGFR TKI resistant) (Experimental): NSCLC participants with previously documented activating EGFR mutation, with any T790M and MET dysregulation status, who received one to three lines of systemic antineoplastic therapy prior to study entry including one line maximum of first or second generation EGFR TKI and who progressed on this EGFR TKI treatment line. Participants were treated at the RP2D of INC280 and EGF816 in fasted state
  Interventions: Drug: Capmatinib; Drug: Nazartinib
- Phase II- Group 2 (EGFRmut, de novo T790M, any MET, 1/3L antineoplastic, EGFR TKI naïve) (Experimental): NSCLC participants harboring T790M mutation in de novo setting, irrespective of the activating mutation status who are treatment naïve or received maximum 2 lines of systemic antineoplastic therapy prior to study entry, but no therapy known to inhibit EGFR. Participants were treated at the RP2D of INC280 and EGF816 in fasted state
  Interventions: Drug: Capmatinib; Drug: Nazartinib
- Phase II- Group 3 (EGFRmut, T790M negative, any MET, 1L antineoplastic) (Experimental): NSCLC participants with previously documented EGFR activating mutation, T790M negative, and any MET status who never received any prior line of systemic antineoplastic systemic therapy prior to study entry. Participants were treated at the RP2D of INC280 and EGF816 in fasted state
  Interventions: Drug: Capmatinib; Drug: Nazartinib
- Phase II- Group 4 (EGFRmut, any T790M, any MET, 1L (treatment naïve) 2-3L antineoplastic) (Experimental): NSCLC participants with previously documented EGFR activating mutations and any T790M and MET status who were treatment naïve or failed maximum 2 prior lines of any systemic antineoplastic therapy for advanced disease. Participants were treated at the RP2D of INC280 and EGF816 in fed state
  Interventions: Drug: Capmatinib; Drug: Nazartinib
- Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L, EGFR TKI resistant) (Experimental): NSCLC participants with previously documented EGFR activating mutation, T790M negative, acquired MET amplification who have progressed on one prior line of therapy for advanced/metastatic NSCLC disease. Participants were to start with INC280 monotherapy (twice a day) and would have had the opportunity to continue to combination of EGF816 (once a day) and INC280 (twice a day) based on radiological disease progression evaluation by investigator's assessment per RECIST 1.1
  Interventions: Drug: Capmatinib; Drug: Nazartinib

INTERVENTIONS:
Drug: Capmatinib — In the Phase 1, capmatinib was administered orally, twice per day, at a dose of 200 mg or 400 mg, in fasted state.
  In the Phase II, participants received capmatinib at the RP2D (400 mg twice per day) in fasted state (Groups 1, 2 and 3) or fed state (Group 4).
  Participants in Phase II Group 5 were to start with capmatinib monotherapy (fasted or fed state) and then would have had the opportunity to continue with the combination of nazartinib and capmatinib (fasted or fed state).
  Other Names: INC280
Drug: Nazartinib — In the Phase 1, nazartinib was administered orally, once a day, at a dose of 50 mg, 75 mg, 100 mg or 150 mg in fasted state.
  In the Phase II, participants received nazartinib at the RP2D (100 mg once daily) in fasted state (Groups 1, 2 and 3) or fed state (Group 4). Participants in Phase II Group 5 were to start with capmatinib monotherapy (fasted or fed state) and then would have had the opportunity to continue with the combination of nazartinib and capmatinib (fasted or fed state).
  Other Names: EGF816

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose (MTD) / recommended phase 2 dose (RP2D) of nazartinib (EGF816) in combination with capmatinib (INC280) and to estimate the preliminary anti-tumor activity of nazartinib in combination with capmatinib in participants with advanced non-small cell lung cancer (NSCLC) with documented EGFR mutation.

DETAILED DESCRIPTION:
This study was designed as a Phase Ib/II, multi-center, open-label study starting with a Phase Ib dose escalation part followed by a Phase II expansion part. Oral nazartinib (once daily) and capmatinib (twice daily) was administered on a continuous schedule until participant experienced unacceptable toxicity, progressive disease (PD) and/or treatment was discontinued at the discretion of the investigator or withdrawal of consent/opposition to use data/biological samples. Study treatment could be continued beyond Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) defined PD, in the judgment of the investigator, when there was evidence of clinical benefit and the subject wished to continue with the study treatment.

In Phase Ib part, participants with NSCLC harboring EGFR activating mutations were enrolled. At the end of the Phase Ib part, once the MTD or RP2D of nazartinib in combination with capmatinib was declared, additional participants with NSCLC were enrolled in the Phase II part in order to assess the preliminary anti-tumor activity of nazartinib in combination with capmatinib. Participants with locally advanced or metastatic NSCLC were assigned into different groups according to their resistance mechanisms.

As per the Protocol amendment 7, an additional group (Group 5) was included into study CINC280X2105C, which was intended to support study CINC280L12301. After thorough and careful assessment of study CINC280L12301 enrollment status, projected study completion timelines, and the changing clinical landscape, Novartis made the decision to discontinue the study. Importantly, this decision was not driven by safety concerns; no new safety signals were observed in the study participants or in the ongoing capmatinib program. As such, Group 5 data was no longer needed and the new arm in study CINC280X2105C was not opened as planned.

ELIGIBILITY:
Key Inclusion criteria:

- Participants in Phase Ib and Phase II Groups 1 to 4: histologically documented, locally advanced or recurrent (stage IIIB who were not eligible for combined modality treatment) or metastatic (Stage IV) NSCLC.

Participants in Phase II Group 5: stage IIIB/IIIC (not amenable to curative surgery, chemoradiation or radiation) or stage IV NSCLC

* Participants in Phase Ib and Phase II Groups 1 to 4: locally documented EGFR mutation L858R and/or ex19del, or a characterized de novo EGFR T790M mutation (or other rare activating mutations that confer sensitivity to 1st and 2nd generation EGFR inhibitors (e.g. L861Q, G719X, S768I), or a characterized de novo EGFRT790M mutation.
* Presence of at least one measurable lesion according to RECIST v.1.1
* ECOG performance status ≤1
* Participants had to be screened for HBV. Participants who were either HBsAg positive or HBV-DNA positive had to be willing and able to take antiviral therapy 1-2 weeks prior to 1st dose of EGF816 treatment and continue on antiviral therapy for at least 4 weeks after the last dose of EGF816.
* Participants had to be screened for HCV. Participants had to have negative hepatitis C antibody (HCV Ab) or were HCV Ab positive but with an undetectable level of HCV-RNA. Note: participants with detectable HCV-RNA were not eligible for the study.
* Phase Ib only: documented progression of disease according to RECIST v1.1 while on continuous treatment with EGFR TKI (e.g.: erlotinib, gefitinib or afatinib).
* Phase II Group 1 (EGFRmut, any T790M, any c-MET, 2/4L antineoplastic, EGFR TKI resistant) only: Participants demonstrated a documented clinical benefit (CR (any duration), PR (any duration), or SD for at least 6 months) on prior EGFR TKI (e.g. erlotinib, gefitinib or afatinib, and subsequently demonstrated progression according to RECIST v1.1.
* Phase II Group 2 (EGFRmut, de novo T790M, any c-MET, 1/3L antineoplastic, EGFR TKI naïve) only: Advanced NSCLC participants who were not previously treated with any therapy known to inhibit EGFR and harbor de novo T790M mutation .
* Phase II Group 3 (EGFRmut, T790M negative, any c-MET, 1L antineoplastic) only: participants had to harbor an EGFR activating mutation and had to be naïve from any line of systemic antineoplastic therapy in the advanced setting.
* Phase II Group 4 (EGFRmut, any T790M, any c-MET, 1L (treatment-naïve), 2//3L antineoplastic): All participants had to harbor an EGFR activating mutation and 2/3L participants had to have failed (defined as intolerance to treatment or documented disease progression) a maximum of 2 prior lines of antineoplastic therapy in the advanced setting
* Phase II Group 5 only: Histologically or cytologically confirmed diagnosis of NSCLC (excluding squamous cell carcinoma) with all the following:

  1. EGFR mutations known to be associated with EGFR TKI sensitivity. This had to be assessed as part of the participant standard of care by a validated test for EGFR mutations, as per local regulations. Exon 19 del, L858R, either alone or in combination with other EGFR sensitivity mutation assessed by a Clinical Laboratory Improvement Amendments (CLIA) certified USA laboratory or an accredited local laboratory outside the USA had to be documented in the participant source documents before the participant consented for pre-screening for MET amplification status.
  2. EGFR T790M negative status for participants who had progressed on first or second generation EGFR TKI, or third generation EGFR TKI other than osimertinib, as per tissue-based result from a CLIA-certified USA laboratory or an accredited local laboratory outside of the USA, by a validated test according to local regulations.
  3. MET gene amplification defined as: Gene copy number (GCN) ≥ 5 per tissue-based result from a CLIA-certified USA laboratory or an accredited local laboratory outside of the USA by a test that is validated according to local regulations with results documented in the participant source documents.
  4. Histological transformation from NSCLC into small cell lung cancer (SCLC) following previous EGFR TKI treatment were excluded.
* Participants had to have progressed on one prior line of therapy either to first/second generation EGFR TKIs, osimertinib or other third generation EGFR TKIs for advanced/metastatic disease (stage IIIB/IIIC [not amenable to curative surgery, chemoradiation or radiation or stage IV NSCLC).
* Participants had to have a life expectancy of at least 3 months.

Key exclusion Criteria:

* Phase Ib:

  * More than one previous treatment line with erlotinib, gefitinib or afatinib
  * Previous treatment with any investigational agent known to inhibit EGFR (mutant or wild-type)
  * Participants who had received more than three prior lines of antineoplastic therapies (including EGFR TKI) in advanced setting.
* Phase II Group 1 (EGFRmut, any T790M, any c-MET, 2/4L antineoplastic, EGFR TKI resistant):

  * More than 3 prior lines of systemic antineoplastic therapies (including EGFR TKI) in the advanced setting
  * More than 1 previous treatment line with 1st or 2nd generation EGFR TKI (e.g. erlotinib, gefitinib, afatinib) in the advanced setting
  * Previous treatment with an investigational or marketed 3rd generation EGFR TKI (e.g. AZD9291, CO-1686, ASP8273, EGF816)
  * Previous treatment with an investigational or marketed agent known to inhibit EGFR (e.g. EGF monoclonal antibody therapy, dual TKI inhibitor).
* Phase II Group 2 (EGFRmut, de novo T790M, any c-MET, 1/3L antineoplastic, EGFR TKI naïve):

  * More than two previous treatment lines of systemic antineoplastic therapies in the advanced setting
  * Previous treatment with an investigational or marketed agent that inhibits EGFR. EGFR inhibitors include (but not limited to) all generations of EGFR TKI (e.g.erlotinib, gefitinib, afatinib, AZD9291, CO-1686, ASP8273, EGF816) or other anti-EGFR or EGFR monoclonal antibody therapy or dual TKI inhibitors.
* Phase II Group 3 (EGFRmut, T790M negative, any c-MET, 1L antineoplastic):

  * De novo EGFR T790M mutation identified by central assessment
  * Previous treatment with any systemic antineoplastic therapy in the advanced setting (NSCLC stage IIIB or IV. Participants who received only one cycle of antineoplastic therapy in the advanced setting were allowed).
* Phase II Group 4 (EGFRmut, any T790M, any c-MET, 1/3L antineoplastic):

  * More than 2 prior lines of systemic antineoplastic therapies in the advanced setting
  * Previous treatment with an investigational or marketed 3rd generation EGFR TKI (e.g. AZD9291, CO-1686, ASP8273, EGF816)
  * Previous treatment with an investigational or marketed agent known to inhibit EGFR (e.g. EGF monoclonal antibody therapy, dual TKI inhibitor).
  * Previous treatment with a c-MET inhibitor or HGF-targeting therapy.
  * Participants with symptomatic brain metastases.
* Phase II Group 5: Participants with symptomatic central nervous system (CNS) metastases who were neurologically unstable or had required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Presence or history of another malignancy. Exception: Participants who had been disease-free for 3 years, or participants with a history of adequately treated in-situ carcinoma of the uterine cervix, completely resected basal or squamous cell carcinoma, non-melanomatous cancer of skin, history of stage IA melanoma that had been cured, were eligible.

For Phase II Group 5: Presence or history of a malignant disease other than NSCLC that had been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.

* Undergone a bone marrow or solid organ transplant.
* Known history of human immunodeficiency virus (HIV) seropositivity (HIV testing is not mandatory).

For Group 5: Participants with known history of testing positive for human immunodeficiency virus (HIV) infection, and with a history of Acquired ImmunoDeficiency Syndrome (AIDS) defining opportunistic infections in the last 12 months prior to the first dose of study treatment had to be excluded

* Participants receiving concomitant immunosuppressive agents or chronic corticosteroids used at the time of study entry except for control of brain metastases, topical applications, inhaled sprays, eye drops or local injections
* Participants with clinically significant, uncontrolled cardiovascular disease
* Presence or history of interstitial lung disease or interstitial pneumonitis
* Participants who had not recovered from all toxicities related to prior anticancer therapies to grade ≤1 (CTCAE v 4.03)
* Participants who had out of range laboratory values
* Participants who received live vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Massachusetts General Hospital Mass General, Boston, Massachusetts, United States
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Edmonton, Alberta, Canada
- Novartis Investigative Site, Marseille, France
- Germany (2):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canarias, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan ROC, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Felip E, Metro G, Soo RA, Wolf J, Solomon BJ, Tan DS, Ardizzoni A, Lee DH, Sequist LV, Barlesi F, Ponce-Aix S, Abreu DR, Campelo MRG, Sprauten M, Djentuh LO, Smith N, Jary A, Belli R, Glaser S, Zou M, Cui X, Giovannini M, Yang JC. Capmatinib plus nazartinib in patients with EGFR-mutated non-small cell lung cancer. Eur J Cancer. 2024 Sep;208:114182. doi: 10.1016/j.ejca.2024.114182. Epub 2024 Jun 22. PMID 38986421
- [Derived] Jia Y, Juarez J, Li J, Manuia M, Niederst MJ, Tompkins C, Timple N, Vaillancourt MT, Pferdekamper AC, Lockerman EL, Li C, Anderson J, Costa C, Liao D, Murphy E, DiDonato M, Bursulaya B, Lelais G, Barretina J, McNeill M, Epple R, Marsilje TH, Pathan N, Engelman JA, Michellys PY, McNamara P, Harris J, Bender S, Kasibhatla S. EGF816 Exerts Anticancer Effects in Non-Small Cell Lung Cancer by Irreversibly and Selectively Targeting Primary and Acquired Activating Mutations in the EGF Receptor. Cancer Res. 2016 Mar 15;76(6):1591-602. doi: 10.1158/0008-5472.CAN-15-2581. Epub 2016 Jan 29. PMID 26825170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 19 investigative sites in 11 countries. Due to early study termination, Group 5 (Phase II part) was never opened
Pre-assignment Details: The screening period began once patients had signed the study informed consent. All screening/baseline evaluations were performed ≤ 28 days before Cycle 1 Day 1.
Groups:
- Phase IB Part- INC280 200mg BID/ EGF816 50mg QD: Combination of INC280 200mg twice daily (BID) and EGF816 50mg once daily (QD) in fasted state in NSCLC participants with previously documented EGFR mutation, who progressed on EGFR TKI treatment
- Phase IB Part- INC280 200mg BID/ EGF816 100mg QD: Combination of INC280 200mg twice daily (BID) and EGF816 100mg once daily (QD) in fasted state in NSCLC participants with previously documented EGFR mutation, who progressed on EGFR TKI treatment
- Phase IB Part- INC280 400mg BID/ EGF816 75mg QD: Combination of INC280 400mg twice daily (BID) and EGF816 75mg once daily (QD) in fasted state in NSCLC participants with previously documented EGFR mutation, who progressed on EGFR TKI treatment
- Phase IB Part- INC280 400mg BID/ EGF816 100mg QD: Combination of INC280 400mg twice daily (BID) and EGF816 100mg once daily (QD) in NSCLC participants with previously documented EGFR mutation, who progressed on EGFR TKI treatment
- Phase IB Part- INC280 400mg BID/ EGF816 150mg QD: Combination of INC280 400mg twice daily (BID) and EGF816 150mg once daily (QD) in fasted state in NSCLC participants with previously documented EGFR mutation, who progressed on EGFR TKI treatment
- Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant): NSCLC participants with previously documented activating EGFR mutation, with any T790M and MET dysregulation status, who received 1 to 3 lines of systemic antineoplastic therapy prior to study entry including one line maximum of 1st or 2nd generation EGFR TKI. Participants were treated with 400 mg twice daily for INC280 and 100 mg once daily for EGF816 in fasted state
- Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve): NSCLC participants harboring T790M mutation in de novo setting, irrespective of the activating mutation status who received none to 2 lines of systemic antineoplastic therapy prior to study entry, but no therapy known to inhibit EGFR. Participants were treated with 400 mg twice daily for INC280 and 100 mg once daily for EGF816 in fasted state
- Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic): NSCLC participants with previously documented EGFR activating mutation, T790M negative, and any MET status who never received any prior line of systemic antineoplastic therapy. Participants were treated with 400 mg twice daily for INC280 and 100 mg once daily for EGF816 in fasted state
- Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic): NSCLC participants with previously documented EGFR activating mutations and any T790M and MET status who received none to 2 prior lines of systemic antineoplastic therapy prior to study entry. Participants were treated with 400 mg twice daily for INC280 and 100 mg once daily for EGF816 in fed state.
- Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant): NSCLC participants with previously documented EGFR activating mutation, T790M negative, acquired MET amplification who have progressed on one prior line of therapy for advanced/metastatic NSCLC disease. Participants started with 400 mg twice daily for INC280 (monotherapy) (fasted or food state) and then had the opportunity to continue with the combination of 400 mg twice daily for INC280 and 100 mg once daily for EGF816 (fasted or food state)
Period: Treatment Phase
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic) | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Started | 4 | 5 | 3 | 16 | 5 | 52 | 3 | 47 | 42 | 0 (Study was early terminated prior to initiating enrollment of Phase II- Group 5)
Completed | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 5 | 6 | 0
Not Completed | 4 | 5 | 3 | 15 | 5 | 50 | 3 | 42 | 36 | 0
Not completed — Progressive Disease | 2 | 5 | 2 | 11 | 4 | 25 | 2 | 30 | 27 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 2 | 1 | 15 | 0 | 5 | 7 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 6 | 1 | 2 | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 0
Not completed — Subject/Guardian Decision | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Period: Post-treatment Follow-up
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic) | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Started | 1 | 0 | 0 | 2 | 0 | 13 | 0 | 5 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 2 | 0 | 13 | 0 | 5 | 3 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 0 | 9 | 0 | 2 | 3 | 0
Not completed — Subject/Guardian Decision | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Phase II-Group 5 arm due to early study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic) | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant) | Total
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5 | 52 | 3 | 47 | 42 | 0 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 2 | 11 | 3 | 33 | 1 | 30 | 24 | 0 | 112
  >=65 years | 1 | 0 | 1 | 5 | 2 | 19 | 2 | 17 | 18 | 0 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 9 | 4 | 38 | 2 | 33 | 24 | 0 | 118
  Male | 0 | 2 | 2 | 7 | 1 | 14 | 1 | 14 | 18 | 0 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 3 | 1 | 10 | 4 | 26 | 2 | 30 | 20 | 0 | 98
  Caucasian | 2 | 2 | 1 | 4 | 1 | 22 | 1 | 16 | 21 | 0 | 70
  Missing | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 8
  Black | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Number of participants with DLTs in the Phase Ib part. A DLT is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 28 days of treatment with EGF816 in combination with INC280 during the escalation part of the study (Phase Ib)
Time Frame: Up to first 28 days of treatment
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816, and who either completed a minimum exposure requirement or who had a DLT during the first 28 days of treatment (Cycle 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 1 | 13 | 5
Participants | 1 | 0 | 0 | 1 | 2

2. Primary Outcome: Phase II Group 1, 2 and 3: Overall Response Rate (ORR) by Investigator's Assessment Per RECIST 1.1
Description: ORR is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) determined by investigator's assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). ORR was assessed in Group 1, 2 and 3 (Phase II part).
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 4 years
Population: All participants in Group 1, 2 or 3 (Phase II part) who received at least one dose of either INC280 or EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47
Percentage of participants | 28.8 [17.1 to 43.10] | 33.3 [0.8 to 90.6] | 61.7 [46.4 to 75.5]

3. Primary Outcome: Phase II Group 4: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: Number of participants in Group 4 (Phase II part) with AEs and SAEs. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Any untoward event resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as SAE.
Time Frame: From start of treatment up to 30 days after last dose of study treatment, assessed up to 3.7 years
Population: All participants in Group 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 42
Participants
  AEs | 42
  SAEs | 26

4. Primary Outcome: Phase II Group 4: Number of Participants With Dose Reductions and Dose Interruptions of INC280 and EGF618
Description: Number of participants with at least one dose reduction of INC280, at least one dose interruption of INC280, at least one dose reduction of EGF816 and at least one dose interruption of EGF816 in the Group 4 (Phase II part).
Time Frame: From start of treatment until end of treatment, assessed up to 3.6 years
Population: All participants in Group 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 42
Participants
  Dose Reduction of INC280 | 30
  Dose Interruption of INC280 | 31
  Dose Reduction of EGF816 | 12
  Dose Interruption of EGF816 | 35

5. Primary Outcome: Phase II Group 4: Dose Intensity
Description: Dose intensity, defined as the ratio of total dose received and actual duration, for participants in Group 4 (Phase II part)
Time Frame: From start of treatment until end of treatment, assessed up to 3.6 years
Population: All participants in Group 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Mean (Standard Deviation); unit: milligram/day
Arm/Group | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 42
milligram/day
  INC280 | 666.2 (148.97)
  EGF816 | 87.4 (14.82)

6. Primary Outcome: Phase II Group 5: ORR Per RECIST 1.1 Based on Investigator's Assessment for INC280 Monotherapy
Description: ORR is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) determined by Investigator assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for participants in Group 5 (Phase II part) while on treatment with INC280 monotherapy.
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 3 years (while on INC280 monotherapy)
Population: Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Arm/Group | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase Ib: Number of Participants With Dose Reductions and Dose Interruptions of INC280 and EGF618
Description: Number of participants in Phase Ib with at least one dose reduction of INC280, at least one dose interruption of INC280, at least one dose reduction of EGF816 and at least one dose interruption of EGF816 .
Time Frame: From start of treatment until end of treatment, assessed up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Count of Participants; unit: Participants
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
Participants
  Dose Reduction of INC280 | 2 | 4 | 2 | 10 | 5
  Dose Interruption of INC280 | 2 | 2 | 2 | 12 | 5
  Dose Reduction of EGF816 | 2 | 1 | 1 | 5 | 3
  Dose Interruption of EGF816 | 2 | 2 | 2 | 11 | 5

8. Secondary Outcome: Phase II Group 1, 2 and 3: Number of Participants With Dose Reductions and Dose Interruptions of INC280 and EGF618
Description: Number of participants in Groups 1, 2 and 3 (Phase II part) with at least one dose reduction of INC280, at least one dose interruption of INC280, at least one dose reduction of EGF816 and at least one dose interruption of EGF816 .
Time Frame: From start of treatment until end of treatment, assessed up to approximately 4 years
Population: All participants in Group 1, 2 and 3 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47
Participants
  Dose Reduction of INC280 | 33 | 3 | 34
  Dose Interruption of INC280 | 31 | 3 | 39
  Dose Reduction of EGF816 | 17 | 2 | 23
  Dose Interruption of EGF816 | 34 | 3 | 40

9. Secondary Outcome: Phase Ib: Dose Intensity
Description: Dose intensity, defined as the ratio of total dose received and actual duration, in Phase Ib participants
Time Frame: From start of treatment until end of treatment, assessed up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Mean (Standard Deviation); unit: milligram/day
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
milligram/day
  INC280 | 319.1 (101.09) | 356.9 (71.14) | 596.3 (200.24) | 658.2 (158.18) | 463.4 (212.52)
  EGF816 | 40.0 (12.60) | 89.6 (17.93) | 60.0 (13.36) | 85.2 (17.28) | 97.7 (36.43)

10. Secondary Outcome: Phase II Group 1, 2 and 3: Dose Intensity
Description: Dose intensity, defined as the ratio of total dose received and actual duration, in Group 1, 2 and 3 (Phase II)
Time Frame: From start of treatment until end of treatment, assessed up to approximately 4 years
Population: All participants in Group 1, 2 and 3 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Mean (Standard Deviation); unit: milligram/day
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47
milligram/day
  INC280 | 662.9 (160.73) | 562.9 (38.36) | 634.7 (172.33)
  EGF816 | 85.2 (18.21) | 76.3 (15.31) | 84.8 (15.53)

11. Secondary Outcome: Phase Ib: Overall Response Rate (ORR) Per RECIST 1.1 Based on Investigator's Assessment
Description: ORR is defined as percentage of participants with best overall response of PR+CR determined by Investigator's assessment in accordance to RECIST 1.1. ORR was assessed in Phase Ib participants.
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
Percentage of participants | 0 [0.0 to 60.2] | 40.0 [5.3 to 85.3] | 33.3 [0.8 to 90.6] | 50.0 [24.7 to 75.3] | 60.0 [14.7 to 94.7]

12. Secondary Outcome: Phase II Group 4: Overall Response Rate (ORR) Per RECIST 1.1 Based on Investigator's Assessment
Description: ORR is defined as percentage of participants with best overall response of PR+CR determined by Investigator's assessment in accordance to RECIST 1.1. ORR was assessed in Group 4 (Phase II) CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 4 years
Population: All participants in Group 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 42
Percentage of participants | 42.9 [27.7 to 59.0]

13. Secondary Outcome: Phase Ib: Progression Free Survival (PFS) Per RECIST 1.1 Based on Investigator's Assessment
Description: PFS is defined as time from date of first dose of study treatment to date of first documented disease progression determined by Investigator assessment in accordance to RECIST 1.1.or death due to any cause. The PFS distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant has not had an event, PFS is censored at the date of last adequate tumor assessment. PFS was assessed in Phase Ib participants
Time Frame: From date of first dose to first documented disease progression or death, assessed up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
Months | 5.6 [3.5 to NA] — NA: Not estimable due to insufficient number of participants with events. | 7.4 [1.6 to NA] — NA: Not estimable due to insufficient number of participants with events. | 3.5 [0.8 to NA] — NA: Not estimable due to insufficient number of participants with events. | 5.7 [1.9 to 42.1] | 14.5 [7.3 to NA] — NA: Not estimable due to insufficient number of participants with events.

14. Secondary Outcome: Phase II Groups 1, 2, 3 and 4: Progression Free Survival (PFS) Per RECIST 1.1 Based on Investigator's Assessment
Description: PFS is defined as time from date of first dose of study treatment to date of first documented disease progression determined by Investigator assessment in accordance to RECIST 1.1.or death due to any cause. The PFS distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant has not had an event, PFS is censored at the date of last adequate tumor assessment. PFS was assessed in Group 1, 2, 3 and 4 (Phase II)
Time Frame: From date of first dose to first documented disease progression or death, assessed up to approximately 4 years
Population: All participants in Group 1, 2 ,3 and 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47 | 42
Months | 5.6 [3.7 to 7.4] | 3.8 [3.7 to NA] — NA: Not estimable due to insufficient number of participants with events. | 10.1 [7.6 to 13.8] | 10.9 [5.6 to 19.2]

15. Secondary Outcome: Phase Ib: Time to Response (TTR) Per RECIST 1.1 Based on Investigator's Assessment
Description: TTR is defined as the time from the date of the first dose to the date of first documented response (CR or PR) determined by Investigator assessment in accordance to RECIST 1.1. The TTR distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant has not had an event, duration was censored at the date of last adequate tumor assessment. TTR was assessed in Phase Ib participants.
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the date of the first dose to the date of first documented response, up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
Months | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — NA: Not estimable due to insufficient number of participants with events. | NA [1.7 to NA] — NA: Not estimable due to insufficient number of participants with events. | 3.5 [1.6 to NA] — NA: Not estimable due to insufficient number of participants with events. | 4.5 [1.9 to NA] — NA: Not estimable due to insufficient number of participants with events.

16. Secondary Outcome: Phase II Groups 1, 2, 3 and 4: Time to Response (TTR) Per RECIST 1.1 Based on Investigator's Assessment
Description: TTR is defined as the time from the date of the first dose to the date of first documented response (CR or PR) determined by Investigator assessment in accordance to RECIST 1.1. The TTR distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant has not had an event, duration was censored at the date of last adequate tumor assessment. TTR was assessed in Group 1, 2, 3 and 4 (Phase II) CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the date of the first dose to the date of first documented response, up to approximately 4 years
Population: All participants in Group 1, 2 ,3 and 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47 | 42
Months | NA [5.4 to NA] — NA: Not estimable due to insufficient number of participants with events. | NA [1.8 to NA] — NA: Not estimable due to insufficient number of participants with events. | 1.9 [1.8 to 5.9] | NA [3.6 to NA] — NA: Not estimable due to insufficient number of participants with events.

17. Secondary Outcome: Phase Ib: Duration of Response (DOR) Per RECIST 1.1 Based on Investigator's Assessment
Description: DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression determined by Investigator assessment in accordance to RECIST 1.1 or death due to underlying cancer. The DOR distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant has not had an event, duration was censored at the date of last adequate tumor assessment. DOR was assessed in Phase Ib participants CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first documented response to first documented disease progression or death, assessed up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816 and had a documented response (CR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 0 | 2 | 1 | 8 | 3
Months |  | 8.8 [5.6 to NA] — NA: Not estimable due to insufficient number of participants with events. | 14.8 [NA to NA] — NA: Not estimable due to insufficient number of participants with events. | 25.3 [3.6 to 47.9] | 8.0 [5.4 to NA] — NA: Not estimable due to insufficient number of participants with events.

18. Secondary Outcome: Phase II Groups 1, 2, 3 and 4: Duration of Response (DOR) Per RECIST 1.1 Based on Investigator's Assessment
Description: DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression determined by Investigator assessment in accordance to RECIST 1.1 or death due to underlying cancer. The DOR distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant has not had an event, duration was censored at the date of last adequate tumor assessment. DOR was assessed in Group 1, 2, 3 and 4 (Phase II) CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first documented response to first documented disease progression or deaths, assessed up to approximately 4 years
Population: All participants in Group 1, 2 ,3 and 4 (Phase II part) who received at least one dose of INC280 or EGF816 and had a documented response (CR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 15 | 1 | 29 | 18
Months | 6.5 [3.7 to 10.8] | 12.0 [NA to NA] — NA: Not estimable due to insufficient number of participants with events. | 11.6 [6.6 to 17.5] | 14.5 [9.2 to NA] — NA: Not estimable due to insufficient number of participants with events.

19. Secondary Outcome: Phase Ib: Disease Control Rate (DCR) Per RECIST 1.1 Based on Investigator's Assessment
Description: DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease (SD) determined by Investigator assessment in accordance to RECIST 1.1. DCR was assessed in Phase Ib participants CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
Time Frame: Up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
Percentage of participants | 100 [39.8 to 100] | 60.0 [14.7 to 94.7] | 33.3 [0.8 to 90.6] | 62.5 [35.4 to 84.8] | 80.0 [28.4 to 99.5]

20. Secondary Outcome: Phase II Group 1, 2 3 and 4: Disease Control Rate (DCR) Per RECIST 1.1 Based on Investigator's Assessment
Description: DCR is defined as the percentage of participants with best overall response of CR, PR, or SD determined by Investigator assessment in accordance to RECIST 1.1. DCR was assessed in Group 1, 2, 3 and 4 (Phase II) CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
Time Frame: Up to approximately 4 years
Population: All participants in Group 1, 2 ,3 and 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47 | 42
Percentage of participants | 59.6 [45.1 to 73.0] | 100 [29.2 to 100] | 93.6 [82.5 to 98.7] | 81.0 [65.9 to 91.4]

21. Secondary Outcome: Phase Ib: Overall Survival (OS)
Description: OS is defined as the time from first dose of the study treatment to the date of death due to any cause. The OS distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant was not known to have died, survival was censored at the date of last contact. OS was assessed in Phase Ib participants
Time Frame: From date of first dose to death, assessed up to approximately 5 years
Population: All participants in Phase Ib part who received at least one dose of INC280 or EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5
Months | 10.1 [8.1 to NA] — NA: Not estimable due to insufficient number of participants with events. | 56.5 [6.5 to NA] — NA: Not estimable due to insufficient number of participants with events. | 7.0 [1.1 to NA] — NA: Not estimable due to insufficient number of participants with events. | 17.2 [5.7 to 58.7] | 31.5 [16.6 to NA] — NA: Not estimable due to insufficient number of participants with events.

22. Secondary Outcome: Phase II Groups 1, 2, 3 and 4: Overall Survival (OS)
Description: OS is defined as the time from first dose of the study treatment to the date of death due to any cause. The OS distribution was estimated using the Kaplan-Meier method and associated 95% confidence intervals were calculated. If a participant was not known to have died, survival was censored at the date of last contact. OS was assessed in Group 1, 2, 3 and 4
Time Frame: From date of first dose to death, assessed up to approximately 4 years
Population: All participants in Group 1, 2 ,3 and 4 (Phase II part) who received at least one dose of INC280 or EGF816
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 52 | 3 | 47 | 42
Months | 18.8 [14.9 to 26.0] | 5.6 [3.7 to NA] — NA: Not estimable due to insufficient number of participants with events. | 25.6 [18.8 to 33.0] | 28.9 [20.5 to NA] — NA: Not estimable due to insufficient number of participants with events.

23. Secondary Outcome: Phase Ib: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 12 Hours (AUC0-12) of INC280
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods.
Time Frame: Pre-dose, 0.5 hours (hr) and 1 hr, 2 hr, 4 hr, 8 hr and 12 hr post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 2 Day 1 (Cycle=28 days)
Population: All participants in Phase Ib part who provided at least one evaluable PK concentration and at least one evaluable PK profile for INC280.
Measure: Mean (Standard Deviation); unit: hours*nanogram/mililiter (hr*ng/mL)
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 1 | 12 | 3
hours*nanogram/mililiter (hr*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 1 | 12 | 3
  Cycle 1 Day 1 | 12300 (4710) | 10500 (4320) | 38300 | 22200 (10700) | 23000 (11600)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 1 | 11 | 2
  Cycle 1 Day 15 | 11600 (3400) | 11800 (3360) | 48800 | 28900 (12700) | 23000 (3440)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 0 | 9 | 2
  Cycle 2 Day 1 | 11300 (4050) | 11100 (1770) |  | 21600 (7370) | 24900 (5190)

24. Secondary Outcome: Phase Ib: Peak Plasma Concentration (Cmax) of INC280
Description: as for outcome 23
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: nanogram/mililiter (ng/mL)
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 1 | 12 | 3
nanogram/mililiter (ng/mL)
  Cycle 1 Day 1 | 3630 (588) | 2530 (1080) | 8000 | 5100 (2550) | 5930 (1330)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 1 | 11 | 2
  Cycle 1 Day 15 | 3070 (1120) | 2840 (1350) | 12000 | 5780 (2640) | 4350 (933)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 0 | 10 | 2
  Cycle 2 Day 1 | 3590 (1620) | 2800 (797) |  | 4830 (1390) | 6370 (1060)

25. Secondary Outcome: Phase Ib: Time to Reach Maximum Concentration (Tmax) of INC280
Description: Pharmacokinetic (PK) parameters were calculated based on INC280 plasma concentrations by using non-compartmental methods. Actual time of sample collection was used (not the nominal time point as per scheduled assessment)
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 1 | 12 | 3
Hours
  Cycle 1 Day 1 | 1.07 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 2.00] | 2.01 [1.00 to 7.67] | 2.00 [1.02 to 2.13]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 1 | 11 | 2
  Cycle 1 Day 15 | 1.12 [1.03 to 2.05] | 2.00 [0.883 to 7.98] | 1.17 [1.17 to 1.17] | 1.97 [0.950 to 4.00] | 1.50 [1.00 to 2.00]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 0 | 10 | 2
  Cycle 2 Day 1 | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 3.83] |  | 1.94 [0.983 to 4.00] | 1.51 [1.02 to 2.00]

26. Secondary Outcome: Phase II Groups 3 and 4: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 12 Hours (AUC0-12) of INC280
Description: as for outcome 23
Time Frame: Pre-dose, 0.5 hours (hr) and 1 hr, 2 hr, 4 hr, 8 hr and 12 hr post-dose on Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle=28 days)
Population: All participants in Group 3 and 4 (Phase II part) who provided at least one evaluable PK concentration and at least one evaluable PK profile for INC280
Measure: Mean (Standard Deviation); unit: hours*nanogram/mililiter (hr*ng/mL)
Arm/Group | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 9 | 15
hours*nanogram/mililiter (hr*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 12
  Cycle 1 Day 1 | 22000 (8000) | 16900 (7360)
  Cycle 2 Day 1: number analyzed (Participants) | 8 | 15
  Cycle 2 Day 1 | 19700 (11200) | 20500 (7440)

27. Secondary Outcome: Phase II Groups 3 and 4: Peak Plasma Concentration (Cmax) of INC280
Description: as for outcome 23
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: nanogram/mililiter (ng/mL)
Arm/Group | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 9 | 15
nanogram/mililiter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 12
  Cycle 1 Day 1 | 4770 (1460) | 3420 (1550)
  Cycle 2 Day 1: number analyzed (Participants) | 8 | 15
  Cycle 2 Day 1 | 4360 (2060) | 3940 (1660)

28. Secondary Outcome: Phase II Groups 3 and 4: Time to Reach Maximum Concentration (Tmax) of INC280
Description: as for outcome 25
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 9 | 15
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 12
  Cycle 1 Day 1 | 1.99 [1.00 to 4.00] | 2.08 [1.85 to 8.00]
  Cycle 2 Day 1: number analyzed (Participants) | 8 | 15
  Cycle 2 Day 1 | 1.47 [1.00 to 7.08] | 3.82 [1.00 to 4.10]

29. Secondary Outcome: Phase Ib: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24) of EGF816
Description: Pharmacokinetic (PK) parameters were calculated based on EGF816 plasma concentrations by using non-compartmental methods.
Time Frame: Pre-dose, 0.5 hours (hr) and 1 hr, 2 hr, 4 hr, 8 hr and 12 hr and 24 hr post-dose on Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 2 Day 1 (Cycle=28 days)
Population: All participants in Phase Ib part who provided at least one evaluable PK concentration and at least one evaluable PK profile for EGF816.
Measure: Mean (Standard Deviation); unit: hours*nanogram/mililiter (hr*ng/mL)
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 13 | 3
hours*nanogram/mililiter (hr*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 2 | 11 | 2
  Cycle 1 Day 1 | 3920 (1450) | 5850 (4380) | 4010 (534) | 5930 (3600) | 10500 (3400)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 5 | 2 | 12 | 2
  Cycle 1 Day 15 | 5200 (2010) | 9630 (4060) | 7330 (108) | 11100 (5340) | 16400 (5670)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 0 | 11 | 2
  Cycle 2 Day 1 | 4080 (1130) | 7460 (2340) |  | 10500 (7480) | 11400 (2360)

30. Secondary Outcome: Phase Ib: Peak Plasma Concentration (Cmax) of EGF816
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nanogram/mililiter (ng/mL)
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 13 | 3
nanogram/mililiter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 5 | 2 | 13 | 3
  Cycle 1 Day 1 | 258 (104) | 465 (323) | 302 (8.49) | 381 (231) | 777 (281)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 3 | 12 | 2
  Cycle 1 Day 15 | 361 (165) | 677 (321) | 517 (180) | 595 (261) | 1010 (354)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 0 | 11 | 2
  Cycle 2 Day 1 | 269 (90.8) | 583 (261) |  | 604 (365) | 814 (137)

31. Secondary Outcome: Phase Ib: Time to Reach Maximum Concentration (Tmax) of EGF816
Description: Pharmacokinetic (PK) parameters were calculated based on EGF816 plasma concentrations by using non-compartmental methods. Actual time of sample collection was used (not the nominal time point as per scheduled assessment)
Time Frame: as for outcome 29
Population: as for outcome 29
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD
Number analyzed (Participants) | 4 | 5 | 3 | 13 | 3
Hours (hr)
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 5 | 2 | 13 | 3
  Cycle 1 Day 1 | 3.03 [1.08 to 4.02] | 3.90 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 8.99] | 4.00 [2.03 to 4.02]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 3 | 12 | 2
  Cycle 1 Day 15 | 2.07 [2.00 to 4.05] | 3.95 [2.00 to 4.00] | 4.00 [2.17 to 4.05] | 5.90 [2.17 to 11.9] | 3.93 [3.83 to 4.02]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 0 | 11 | 2
  Cycle 2 Day 1 | 4.00 [3.95 to 4.00] | 4.00 [2.00 to 4.00] |  | 4.00 [1.98 to 7.00] | 3.05 [2.10 to 4.00]

32. Secondary Outcome: Phase II Groups 3 and 4: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24) of EGF816
Description: as for outcome 29
Time Frame: Pre-dose, 0.5 hours (hr) and 1 hr, 2 hr, 4 hr, 8 hr and 12 hr and 24 hr post-dose on Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle=28 days)
Population: All participants in Group 3 and 4 (Phase II part) who provided at least one evaluable PK concentration and at least one evaluable PK profile for EGF816.
Measure: Mean (Standard Deviation); unit: hours*nanogram/mililiter (hr*ng/mL)
Arm/Group | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 7 | 15
hours*nanogram/mililiter (hr*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 12
  Cycle 1 Day 1 | 6390 (2460) | 3420 (1700)
  Cycle 2 Day 1: number analyzed (Participants) | 5 | 15
  Cycle 2 Day 1 | 11100 (2000) | 7670 (3330)

33. Secondary Outcome: Phase II Groups 3 and 4: Peak Plasma Concentration (Cmax) of EGF816
Description: as for outcome 29
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: nanogram/mililiter (ng/mL)
Arm/Group | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 7 | 15
nanogram/mililiter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 12
  Cycle 1 Day 1 | 448 (184) | 239 (107)
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 15
  Cycle 2 Day 1 | 658 (117) | 447 (175)

34. Secondary Outcome: Phase II Groups 3 and 4: Time to Reach Maximum Concentration (Tmax) of EGF816
Description: as for outcome 31
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic)
Number analyzed (Participants) | 7 | 15
Hours (hr)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 12
  Cycle 1 Day 1 | 4.00 [1.12 to 8.00] | 4.00 [1.85 to 8.00]
  Cycle 2 Day 1: number analyzed (Participants) | 6 | 15
  Cycle 2 Day 1 | 4.00 [2.00 to 4.13] | 4.00 [3.82 to 8.00]

35. Secondary Outcome: Phase II Group 5: Duration of Response (DOR) Per RECIST 1.1 Based on Investigator's Assessment for INC280 Monotherapy
Description: DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1 for participants in Group 5 (Phase II) while on INC280 monotherapy treatment.
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first documented response to the date of first documented disease progression or death, assessed up to approximately 3 years (while on INC280 monotherapy)
Population: Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Arm/Group | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 0

36. Secondary Outcome: Phase II Group 5: Disease Control Rate (DCR) Per RECIST 1.1 Based on Investigator's Assessment for INC280 Monotherapy
Description: DCR is defined as the percentage of participants with best overall response of CR, PR, or SD determined by Investigator assessment in accordance to RECIST 1.1 for participants in Group 5 (Phase II) while on INC280 monotherapy treatment.
  CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
Time Frame: Up to approximately 3 years (while on INC280 monotherapy)
Population: Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Arm/Group | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 0

37. Secondary Outcome: Phase II Group 5: Progression Free Survival (PFS) Per RECIST 1.1 Based on Investigator's Assessment for INC280 Monotherapy
Description: PFS is defined as time from date of first dose of study treatment to date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1 for participants in Group 5 (Phase II) while on INC280 monotherapy treatment.
Time Frame: Up to approximately 3 years (while on INC280 monotherapy)
Population: Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Arm/Group | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 0

38. Secondary Outcome: Phase II Group 5: Number of Participants With Dose Modifications for INC280 Monotherapy as Well as INC280 in Combination With EGF816 Therapy
Description: Number of participants with dose modifications for INC280 monotherapy as well as INC280 in combination with EGF816 therapy
Time Frame: From start of treatment until end of treatment, up to approximately 3 years
Population: Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Arm/Group | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 0

39. Secondary Outcome: Phase II Group 5: Dose Intensity for INC280 Monotherapy as Well as INC280 in Combination With EGF816 Therapy
Description: Dose intensity is defined as the ratio of total dose received and actual duration for INC280 monotherapy as well as INC280 in combination with EGF816 therapy in Group 5 (Phase II)
Time Frame: From start of treatment until end of treatment, up to approximately 3 years
Population: Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Arm/Group | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 0

40. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study medication to 30 days after the last dose of study medication.
  Post-treatment survival follow-up deaths were collected after 30 days post-treatment.
  All deaths refer to the sum of on-treatment and post-treatment deaths
Time Frame: On-treatment: up to approximately 5 years (Phase Ib) and 4 years (Phase II). Post-treatment survival follow-up: Up to approximately 5 years (Phase Ib) and 4 years (Phase II).
Population: All participants in Phase Ib part and Group 1, 2, 3 and 4 (Phase II part) who received at least one dose of INC280 or EGF816. Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD | Phase II- Group 1 (EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant) | Phase II- Group 2 (EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve) | Phase II- Group 3 (EGFRmut, T790M Negative, Any MET, 1L Antineoplastic) | Phase II- Group 4 (EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic) | Phase II- Group 5 (EGFRmut, T790M-, MET GCN≥5, 2L Antineoplastic, EGFR TKI Resistant)
Number analyzed (Participants) | 4 | 5 | 3 | 16 | 5 | 52 | 3 | 47 | 42 | 0
Participants
  On-treatment deaths | 0 | 0 | 1 | 2 | 0 | 9 | 2 | 5 | 1 |
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 4 | 3 | 2 | 13 | 5 | 40 | 1 | 37 | 33 | 0
  Post-treatment survival follow-up deaths | 4 | 3 | 2 | 9 | 3 | 26 | 1 | 25 | 22 |
  All deaths | 4 | 3 | 3 | 11 | 3 | 35 | 3 | 30 | 23 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose of study treatment, up to approx. 5 years (Phase Ib) and 4 years (Phase II). Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approx. 5 years (Phase Ib) and 4 years (Phase II).These are not considered AEs
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
  Due to early termination of the study, no participants were enrolled in Group 5 (Phase II part)
Groups:
- Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (On-treatment); Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (On-treatment); Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (On-treatment); Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (On-treatment); Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (On-treatment); Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (On-treatment); Phase II- EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (On-treatment); Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (On-treatment); Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (On-treatment): AEs collected during on-treatment period (up to 30 days post-treatment)
- Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (Post-treatment FU); Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (Post-treatment FU); Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (Post-treatment FU); Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (Post-treatment FU); Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (Post-treatment FU); Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (Post-treatment FU); Phase II-EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (Post-treatment FU); Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (Post-treatment FU); Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (Post-treatment FU): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (On-treatment) | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (Post-treatment FU) | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (On-treatment) | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (Post-treatment FU) | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (On-treatment) | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (Post-treatment FU) | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (On-treatment) | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (Post-treatment FU) | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (On-treatment) | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (Post-treatment FU) | Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (On-treatment) | Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (Post-treatment FU) | Phase II- EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (On-treatment) | Phase II-EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (Post-treatment FU) | Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (On-treatment) | Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (Post-treatment FU) | Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (On-treatment) | Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (Post-treatment FU)
All-Cause Mortality (participants affected / at risk) | 0/4 | 4/4 | 0/5 | 3/3 | 1/3 | 2/2 | 2/16 | 9/13 | 0/5 | 3/5 | 9/52 | 26/40 | 2/3 | 1/1 | 5/47 | 25/37 | 1/42 | 22/33
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/0 | 2/5 | 0/0 | 3/3 | 0/0 | 11/16 | 0/0 | 4/5 | 0/0 | 29/52 | 0/0 | 2/3 | 0/0 | 33/47 | 0/0 | 26/42 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 5/5 | 0/0 | 3/3 | 0/0 | 16/16 | 0/0 | 5/5 | 0/0 | 51/52 | 0/0 | 3/3 | 0/0 | 47/47 | 0/0 | 42/42 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (On-treatment) (N=4) | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (On-treatment) (N=5) | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (On-treatment) (N=3) | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (On-treatment) (N=16) | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (On-treatment) (N=5) | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (Post-treatment FU) (N=0) | Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (On-treatment) (N=52) | Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (Post-treatment FU) (N=0) | Phase II- EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (On-treatment) (N=3) | Phase II-EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (Post-treatment FU) (N=0) | Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (On-treatment) (N=47) | Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (Post-treatment FU) (N=0) | Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (On-treatment) (N=42) | Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (Post-treatment FU) (N=0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Cardiac arrest (Cardiac disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Myocardial ischaemia (Cardiac disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Pericardial effusion (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Visual impairment (Eye disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Ascites (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Colitis (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Constipation (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Diarrhoea (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Hiatus hernia (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Inguinal hernia (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Nausea (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA
Vomiting (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Asthenia (General disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Fatigue (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 1 | NA | 1 | NA
General physical health deterioration (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Influenza like illness (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Non-cardiac chest pain (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Oedema (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Pyrexia (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 4 | NA | 2 | NA
Hepatic failure (Hepatobiliary disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Anaphylactic shock (Immune system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Hypersensitivity (Immune system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 1 | NA
Cellulitis (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA | 1 | NA | 0 | NA | 2 | NA | 3 | NA
Empyema (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Enterocolitis infectious (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Erysipelas (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Herpes zoster (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Herpes zoster meningitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Influenza (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Lower respiratory tract infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Meningitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Meningitis aseptic (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Necrotising fasciitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Pleural infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Pneumonia (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 5 | NA | 0 | NA | 0 | NA | 4 | NA
Pneumonia aspiration (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Pneumonia chlamydial (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Respiratory tract infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Sepsis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Soft tissue infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Urinary tract infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Urosepsis (Infections and infestations) | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Fall (Injury, poisoning and procedural complications) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Alanine aminotransferase increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Amylase increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Aspartate aminotransferase increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Blood bilirubin increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Blood creatinine increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Ejection fraction decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Neutrophil count decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Weight decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 0 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Aphasia (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Brain oedema (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Cerebral ischaemia (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Dysarthria (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Epilepsy (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Headache (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 0 | NA
Hydrocephalus (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Hypertensive hydrocephalus (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Loss of consciousness (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Neurological decompensation (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Seizure (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 1 | NA | 2 | NA | 0 | NA | 1 | NA | 1 | NA
Speech disorder (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Spinal cord compression (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Tremor (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Wernicke's encephalopathy (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Apathy (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Confusional state (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Renal failure (Renal and urinary disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 1 | NA | 2 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 3 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 4 | NA | 3 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 1 | NA | 1 | NA | 1 | NA | 1 | NA | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 3 | NA | 0 | NA
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Purpura (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Rash macular (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 4 | NA | 0 | NA | 0 | NA | 1 | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Embolism (Vascular disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Hypertensive crisis (Vascular disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Hypotension (Vascular disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (On-treatment) (N=4) | Phase IB Part- INC280 200mg BID/ EGF816 50mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (On-treatment) (N=5) | Phase IB Part- INC280 200mg BID/ EGF816 100mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (On-treatment) (N=3) | Phase IB Part- INC280 400mg BID/ EGF816 75mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (On-treatment) (N=16) | Phase IB Part- INC280 400mg BID/ EGF816 100mg QD (Post-treatment FU) (N=0) | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (On-treatment) (N=5) | Phase IB Part- INC280 400mg BID/ EGF816 150mg QD (Post-treatment FU) (N=0) | Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (On-treatment) (N=52) | Phase II- EGFRmut, Any T790M, Any MET, 2/4L Antineoplastic, EGFR TKI Resistant (Post-treatment FU) (N=0) | Phase II- EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (On-treatment) (N=3) | Phase II-EGFRmut, de Novo T790M, Any MET, 1/3L Antineoplastic, EGFR TKI naïve (Post-treatment FU) (N=0) | Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (On-treatment) (N=47) | Phase II- EGFRmut, T790M Negative, Any MET, 1L Antineoplastic (Post-treatment FU) (N=0) | Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (On-treatment) (N=42) | Phase II-EGFRmut, Any T790M, Any MET, 1/3L Antineoplastic (Post-treatment FU) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 2 | NA | 2 | NA | 1 | NA | 9 | NA | 1 | NA | 11 | NA | 4 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 3 | NA | 0 | NA | 1 | NA | 1 | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | NA | 2 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 4 | NA | 0 | NA | 3 | NA | 2 | NA
Angina pectoris (Cardiac disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 1 | NA
Bradycardia (Cardiac disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Deafness (Ear and labyrinth disorders) | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Deafness transitory (Ear and labyrinth disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Ear pain (Ear and labyrinth disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 0 | NA | 3 | NA | 3 | NA
Tinnitus (Ear and labyrinth disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 6 | NA | 0 | NA
Hyperthyroidism (Endocrine disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Eye pruritus (Eye disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 1 | NA
Eye swelling (Eye disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Eyelid oedema (Eye disorders) | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Vision blurred (Eye disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Vitreous floaters (Eye disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 3 | NA
Abdominal distension (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 7 | NA | 4 | NA
Abdominal pain (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 4 | NA | 0 | NA | 5 | NA | 2 | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 4 | NA | 0 | NA | 6 | NA | 7 | NA
Constipation (Gastrointestinal disorders) | 1 | NA | 0 | NA | 1 | NA | 5 | NA | 2 | NA | 4 | NA | 1 | NA | 6 | NA | 8 | NA
Diarrhoea (Gastrointestinal disorders) | 1 | NA | 1 | NA | 1 | NA | 6 | NA | 2 | NA | 20 | NA | 2 | NA | 26 | NA | 20 | NA
Dry mouth (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 0 | NA | 1 | NA | 3 | NA
Dyspepsia (Gastrointestinal disorders) | 0 | NA | 0 | NA | 1 | NA | 4 | NA | 0 | NA | 10 | NA | 0 | NA | 9 | NA | 6 | NA
Dysphagia (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 3 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 1 | NA | 2 | NA | 6 | NA
Lip blister (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Lip dry (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Mouth ulceration (Gastrointestinal disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 4 | NA | 4 | NA
Nausea (Gastrointestinal disorders) | 2 | NA | 0 | NA | 2 | NA | 11 | NA | 5 | NA | 28 | NA | 3 | NA | 27 | NA | 19 | NA
Odynophagia (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Stomatitis (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 2 | NA | 5 | NA | 0 | NA | 12 | NA | 3 | NA
Toothache (Gastrointestinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 0 | NA
Vomiting (Gastrointestinal disorders) | 0 | NA | 0 | NA | 1 | NA | 6 | NA | 3 | NA | 20 | NA | 1 | NA | 22 | NA | 11 | NA
Asthenia (General disorders) | 2 | NA | 2 | NA | 1 | NA | 4 | NA | 0 | NA | 6 | NA | 1 | NA | 18 | NA | 10 | NA
Chest pain (General disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Chills (General disorders) | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 0 | NA | 2 | NA | 0 | NA
Face oedema (General disorders) | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 1 | NA | 2 | NA | 0 | NA | 2 | NA | 1 | NA
Fatigue (General disorders) | 2 | NA | 0 | NA | 2 | NA | 6 | NA | 2 | NA | 14 | NA | 2 | NA | 9 | NA | 9 | NA
Gait disturbance (General disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Influenza like illness (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 2 | NA | 5 | NA
Non-cardiac chest pain (General disorders) | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 8 | NA | 1 | NA | 6 | NA | 6 | NA
Oedema peripheral (General disorders) | 1 | NA | 1 | NA | 2 | NA | 8 | NA | 4 | NA | 27 | NA | 3 | NA | 31 | NA | 26 | NA
Pain (General disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 2 | NA | 1 | NA
Peripheral swelling (General disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 3 | NA
Pyrexia (General disorders) | 1 | NA | 1 | NA | 0 | NA | 7 | NA | 3 | NA | 8 | NA | 0 | NA | 11 | NA | 12 | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 1 | NA
Anaphylactoid reaction (Immune system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Hypersensitivity (Immune system disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Bronchitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 0 | NA | 2 | NA | 2 | NA
Cellulitis (Infections and infestations) | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 3 | NA | 5 | NA
Conjunctivitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 0 | NA | 1 | NA
Cystitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA
Folliculitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 1 | NA
Gastroenteritis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA
Herpes zoster (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 3 | NA
Infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Nasopharyngitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 5 | NA | 0 | NA | 5 | NA | 5 | NA
Paronychia (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA | 5 | NA | 2 | NA | 3 | NA | 0 | NA | 7 | NA | 7 | NA
Pharyngitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA
Pneumonia (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 2 | NA | 0 | NA | 2 | NA | 2 | NA
Respiratory tract infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 0 | NA
Rhinitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 1 | NA | 2 | NA | 1 | NA
Sinobronchitis (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Skin infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA
Tooth infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Upper respiratory tract infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 4 | NA | 0 | NA | 9 | NA | 0 | NA | 6 | NA | 6 | NA
Urinary tract infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 5 | NA | 0 | NA | 4 | NA | 8 | NA
Viral infection (Infections and infestations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Alanine aminotransferase increased (Investigations) | 2 | NA | 0 | NA | 0 | NA | 2 | NA | 2 | NA | 7 | NA | 2 | NA | 13 | NA | 13 | NA
Amylase increased (Investigations) | 2 | NA | 2 | NA | 1 | NA | 8 | NA | 2 | NA | 11 | NA | 1 | NA | 11 | NA | 7 | NA
Aspartate aminotransferase increased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 4 | NA | 2 | NA | 13 | NA | 11 | NA
Blood albumin decreased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Blood alkaline phosphatase increased (Investigations) | 1 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 6 | NA | 2 | NA
Blood bilirubin increased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 1 | NA
Blood creatine increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Blood creatine phosphokinase increased (Investigations) | 0 | NA | 1 | NA | 1 | NA | 4 | NA | 0 | NA | 5 | NA | 0 | NA | 5 | NA | 6 | NA
Blood creatinine increased (Investigations) | 2 | NA | 2 | NA | 0 | NA | 8 | NA | 2 | NA | 10 | NA | 1 | NA | 16 | NA | 15 | NA
Blood glucose increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Blood potassium increased (Investigations) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Blood triglycerides increased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Blood urea increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 2 | NA
Blood uric acid increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 0 | NA
C-reactive protein increased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Electrocardiogram QT prolonged (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 1 | NA | 3 | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 2 | NA | 0 | NA | 5 | NA | 5 | NA
Haemoglobin decreased (Investigations) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Lipase increased (Investigations) | 0 | NA | 1 | NA | 0 | NA | 4 | NA | 1 | NA | 12 | NA | 0 | NA | 7 | NA | 8 | NA
Lymphocyte count decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Protein total decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 4 | NA | 0 | NA | 0 | NA | 3 | NA
Weight decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 2 | NA
Weight increased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 2 | NA | 3 | NA | 0 | NA | 4 | NA | 2 | NA
White blood cell count decreased (Investigations) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | NA | 0 | NA | 0 | NA | 10 | NA | 1 | NA | 14 | NA | 1 | NA | 14 | NA | 9 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 2 | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 3 | NA | 0 | NA | 0 | NA | 1 | NA
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 1 | NA | 5 | NA | 1 | NA | 9 | NA | 0 | NA | 10 | NA | 7 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 2 | NA | 0 | NA | 3 | NA | 0 | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 5 | NA | 1 | NA | 4 | NA | 2 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 1 | NA | 4 | NA | 1 | NA | 3 | NA | 3 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 3 | NA | 0 | NA | 4 | NA | 0 | NA | 1 | NA | 2 | NA
Hypophagia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 2 | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | NA | 1 | NA | 1 | NA | 2 | NA | 1 | NA | 3 | NA | 0 | NA | 10 | NA | 6 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 7 | NA | 8 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 3 | NA | 1 | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 2 | NA | 4 | NA | 0 | NA | 12 | NA | 14 | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 3 | NA | 2 | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 4 | NA | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | NA | 1 | NA | 2 | NA | 1 | NA | 2 | NA | 0 | NA | 3 | NA | 0 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 3 | NA | 4 | NA | 0 | NA | 7 | NA | 7 | NA
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Amnesia (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Dizziness (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 4 | NA | 1 | NA | 9 | NA | 0 | NA | 11 | NA | 10 | NA
Dysaesthesia (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Dysgeusia (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 4 | NA | 1 | NA
Epilepsy (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Headache (Nervous system disorders) | 0 | NA | 1 | NA | 0 | NA | 7 | NA | 0 | NA | 7 | NA | 1 | NA | 17 | NA | 12 | NA
Hypoaesthesia (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 1 | NA | 0 | NA | 3 | NA | 2 | NA
Lethargy (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA
Neuropathy peripheral (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Post herpetic neuralgia (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Seizure (Nervous system disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 1 | NA | 3 | NA | 1 | NA
Syncope (Nervous system disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Anxiety (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 4 | NA | 0 | NA
Confusional state (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Depression (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA
Insomnia (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 4 | NA | 0 | NA | 3 | NA | 4 | NA
Sleep disorder (Psychiatric disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Hypertonic bladder (Renal and urinary disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Renal failure (Renal and urinary disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Perineal pain (Reproductive system and breast disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Prostatomegaly (Reproductive system and breast disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 2 | NA | 2 | NA | 5 | NA | 1 | NA | 10 | NA | 1 | NA | 11 | NA | 14 | NA
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 1 | NA | 1 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 1 | NA | 1 | NA | 4 | NA | 1 | NA | 11 | NA | 1 | NA | 13 | NA | 7 | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 4 | NA | 0 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 2 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 4 | NA | 0 | NA | 0 | NA | 0 | NA
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 5 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 3 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 0 | NA | 1 | NA | 3 | NA | 0 | NA | 2 | NA | 0 | NA | 2 | NA | 5 | NA
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Acne (Skin and subcutaneous tissue disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 1 | NA | 2 | NA | 0 | NA | 0 | NA | 0 | NA | 4 | NA | 0 | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 2 | NA | 2 | NA | 2 | NA | 0 | NA | 10 | NA | 4 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 5 | NA | 1 | NA | 5 | NA | 0 | NA | 7 | NA | 5 | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 0 | NA | 1 | NA | 6 | NA
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 0 | NA | 5 | NA | 1 | NA | 6 | NA | 0 | NA | 9 | NA | 14 | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 7 | NA | 0 | NA | 11 | NA | 9 | NA
Rash macular (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | NA | 1 | NA | 1 | NA | 1 | NA | 0 | NA | 1 | NA | 3 | NA | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | NA | 2 | NA | 0 | NA | 3 | NA | 4 | NA | 10 | NA | 1 | NA | 14 | NA | 9 | NA
Rash papular (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 2 | NA | 2 | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA | 1 | NA | 0 | NA | 3 | NA | 1 | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 2 | NA
Hot flush (Vascular disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 0 | NA
Hypotension (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 2 | NA | 1 | NA | 1 | NA | 4 | NA | 1 | NA
Pallor (Vascular disorders) | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA
Thrombosis (Vascular disorders) | 0 | NA | 0 | NA | 0 | NA | 1 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02335944/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02335944/SAP_001.pdf